CLINICAL TRIAL: NCT00888836
Title: Prospective Randomized Controlled Trial on the Effect of Gastric Bypass and Biliopancreatic Diversion on Type 2 Diabetes Mellitus in Patients With BMI > 35 vs. Medical Therapy
Brief Title: Diet and Medical Therapy Versus Bariatric Surgery in Type 2 Diabetes
Acronym: DIBASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Assistant Professor of Internal Medicine, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSC-2009-1
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
Keywords: bariatric surgery; GBP; BPD; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GBP (Active Comparator): Type 2 diabetic subjects with BMI ≥ 35, poor glycemic control (HbA1c ≥ 7.0%) and diabetes duration ≥ 5 years undergo gastric bypass
  Interventions: Procedure: Bariatric surgery: Gastric bypass
- BPD 2 (Active Comparator): Type 2 diabetic subjects with BMI ≥ 35, poor glycemic control (HbA1c ≥ 7.0%) and diabetes duration ≥ 5 years undergo bilio-pancreatic diversion
  Interventions: Procedure: Bariatric surgery: Bilio-pancreatic diversion
- Med Ter3 (Active Comparator): Type 2 diabetic subjects with BMI ≥ 35, poor glycemic control (HbA1c ≥ 7.0%) and diabetes duration ≥ 5 yearsundergo medical therapy
  Interventions: Behavioral: anti-diabetic drugs and behavioral suggestions

INTERVENTIONS:
Procedure: Bariatric surgery: Gastric bypass — Gastric bypass (GBP): A subcardial gastric pouch with a 30±10 ml capacity will be created on a naso-gastric 36F calibrating tube by sectioning the stomach with a linear stapler 3-4 cm horizontally on the lesser curve, 4 cm distal to the e-g junction, and then vertically until attainment of the angle of Hiss. After identification of the Treitz ligament, the jejunum will be transected at 100 cm from the ligament of Treitz and the two stumps will be closed. The distal stump will be anastomosed to the distal end of the gastric pouch. The preferred gastro-jejunal anastomosis is the totally hand-sewn one, but it can be performed using any other the technique the surgeon is more familiar with. Finally, the proximal stump of the transacted bowel will be joined end-to-side to the jejunum 150 cm distal to the gastroenterostomy.
  Arms: GBP
Procedure: Bariatric surgery: Bilio-pancreatic diversion — Biliopancreatic diversion (BPD): A distal two-third gastrectomy will be carried out aiming at leaving an about 400 ml gastric remnant. The gastrointestinal continuity will be re-established by sectioning the small bowel 300 cm proximal to the ileocecal valve, closing the intestinal stumps, and joining the proximal one end-to-side to the distal ileum at 50 cm from the ligament of Treitz. The distal stump of the transacted bowel will be anastomosed to the left corner of the gastric stump, preferably in a totally hand-sewn fashion.
  Arms: BPD 2
Behavioral: anti-diabetic drugs and behavioral suggestions — Medical therapies (oral hypoglycemic agents and insulin) are optimized on an individual basis. Lifestyle modification programs, including reduced energy and fat (<30% total fat and <10% saturated fat, high fibre content) intake and increased physical exercise (suggested at least 30 minutes of brisk walking every day possibly associated with a moderate intensity aerobic activity twice a week), are tailor made by an experienced diabetologist assisted by a dietitian. After the two years, the patients in control group will be offered the choice to undergo one of the two surgical procedures.
  Arms: Med Ter3

SUMMARY:
It is generally held that ß-cell function is irreversibly lost already at the time the disease manifests itself and thereafter continues to decline linearly with time. Several studies, however, have documented the possibility that ß-cell function may be restored, at least partially, in type 2 diabetes. Of major relevance to the issue of ß-cell recovery in diabetes are the following findings:

* bariatric surgery in morbidly obese patients with type 2 diabetes can restore euglycaemia, the acute insulin response to glucose and insulin sensitivity;
* recent studies have reported that diabetic subjects return to euglycaemia and normal insulin levels within days after surgery, long before a significant weight loss has occurred; and
* whereas gastric bypass (GBP) improves insulin sensitivity in proportion to weight loss, bilio-pancreatic diversion (BPD) improves insulin action out of proportion to weight loss, i.e., it normalizes it at a time when patients are still markedly obese. Because RYGB is a predominantly restrictive procedure involving the foregut, whereas BPD is a predominantly malabsorptive procedure involving the distal gastro-intestinal (GI) tract, these findings suggest that the control of both insulin action and ß-cell function is influenced by signals originating from the GI tract.

The principal aim of this study is to verify the effect on type 2 diabetes mellitus (T2DM) of GBP and BPD, the two operations which have shown specific actions on glucose homeostasis control, in type 2 diabetic patients with BMI > 35 kg/m2, and to compare this effect with matched T2DM control patients receiving the standard of medical care.

DETAILED DESCRIPTION:
ß-cell dysfunction and insulin resistance are the main pathophysiological defects responsible for the development of hyperglycaemia [1]. Both these defects predict incident diabetes in high-risk subjects [2]. Insulin resistance per se is not sufficient to cause hyperglycaemia; mild degrees of ß-cell dysfunction, on the other hand, may not result in diabetic hyperglycaemia in insulin sensitive individuals. It is only when impaired ß-cell function occurs in the background of insulin resistance that plasma glucose levels begin to rise (as is the case of individuals with impaired glucose tolerance [3]). The occurrence of postprandial, or day-long, hyperglycaemia further compromises both ß-cell function and insulin action, a phenomenon called glucose toxicity [4-6]. As a consequence, the vast majority of patients with established type 2 diabetes present, in addition to marked insulin resistance, a clear defect in ß-cell function, which is generally proportional to the severity of the hyperglycaemia [7]. Of note is that the extent of ß-cell dysfunction in type 2 patients may be misjudged when ß-cell function is inferred from simple measurements of fasting or postprandial plasma insulin concentrations. In fact, insulin secretion increases (in non-linear manner [8]) in insulin resistant individuals, a compensatory response aimed at maintaining glucose tolerance. As a consequence, the absolute insulin hypersecretion (particularly in the fasting state) commonly found in patients with IGT or diabetes masks the underlying defect in the ability of the ß-cell to cope with nutrient stimulation.

It is generally held that ß-cell function is irreversibly lost already at the time the disease manifests itself and thereafter continues to decline linearly with time. Several studies, however, have documented the possibility that ß-cell function may be restored, at least partially, in type 2 diabetes [9-13]. Of major relevance to the issue of ß-cell recovery in diabetes are the following findings: (a) bariatric surgery in morbidly obese patients with type 2 diabetes can restore euglycaemia, the acute insulin response to glucose [14-17] and insulin sensitivity [18,19]; (b) recent studies have reported that diabetic subjects return to euglycaemia and normal insulin levels within days after surgery, long before a significant weight loss has occurred [20]; and (c) whereas RYGB improves insulin sensitivity in proportion to weight loss, BPD improves insulin action out of proportion to weight loss, i.e., it normalises it at a time when patients are still markedly obese [21]. Because RYGB is a predominantly restrictive procedure involving the foregut whereas BPD is a predominantly malabsorptive procedure involving the distal GI tract, these findings suggest that the control of both insulin action and ß-cell function is influenced by signals originating from the GI tract.

Some studies have investigated the hormonal changes that follow bariatric surgery. In most cases, however, clinical testing was performed after significant weight reduction, thereby making it difficult to establish whether any observed hormonal effect was the cause or the consequence of weight loss and diabetes resolution. Recently, it has been reported that RYGB induces rapid normalisation of blood glucose and insulin levels in concomitance with significant changes of the levels of hormones involved in the regulation of glucose metabolism (ACTH, leptin and GIP) in the early postoperative period [22]. It has been proposed that the incretins could be one of the key mediators of the anti-diabetic effects of certain types of bariatric surgery. Previous data have shown that the significant weight loss observed after various bariatric procedures was accompanied by improvement of diabetes control and increased GLP-1 levels. However, most studies were cross sectional [23,24], reported fasting [25] rather than post-prandial GLP-1 levels, and compared various types of surgery such as jejuno-ileal bypass (JIB) [26,27] or bilio-pancreatic diversion (BPD) [27], often leading to inconclusive results. Data on fasting GIP levels after bariatric surgery are inconsistent, reporting either a decrease [25,28,29] or an increase [23,24]. GLP-1 levels increase after a meal in patients after RY-GBP [30] or with oral glucose after BPD [30]. Meal-stimulated GIP levels have been reported to increase after JIB [23], or to decrease after GBP, JIB or BPD surgery [26,29,31,32]. None of these studies, however, measured GLP-1 and GIP simultaneously, reported the incretin levels and effect on insulin secretion (with the exception of the last quoted one, which reported both GIP and insulin response to meal markedly reduced after BPD), or was done in diabetic patients.

Some authors have suggested that an enhanced release of GLP-1, triggered by the earlier presentation of undigested food to lower segments of the bowel, might be involved in the glycaemic improvement consequent to bypass procedures for obesity surgery.

Collectively, these observations clearly suggest that there is a large margin for ß-cell recovery of function in type 2 diabetes and that different segments of the gut participate differentially in such recovery.

The primary end-points of the study are the differences in the proportions of patients reaching partial or complete remission of type 2 diabetes between conventional therapy and BPD or conventional therapy and RYGB.

In particular, according to Buse et al (Diabetes Care 2009; 32:2133-35) partial remission is defined as fasting glucose values of 100-125 mg/dl [5.6-6.9 mmol/l]) and HbA1c<6.5%, of at least 1 year's duration in the absence of active pharmacologic therapy. Complete remission is referred to fasting glucose <100 mg/dl [5.6 mmol/l]) and HbA1c in the normal range of at least 1 year's duration in the absence of active pharmacologic therapy.

Secondary endpoints Secondary endpoints include percentage change of fasting plasma glucose levels, glycated hemoglobin, weight, waist circumference, blood pressure, cholesterol, HDL-cholesterol and triglycerides, and hard cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes and BMI ≥35 kg.m-2
* age between 30 and 60 years
* duration of diabetes ≥ 5 years
* poor glycemic control (i.e., HbA1c ≥ 7.0%) in spite a medical antidiabetic therapy in accordance with good clinical practice (GCP)

Exclusion Criteria:

* pregnancy
* medical conditions requiring acute hospitalisation
* severe diabetes complications or associated medical conditions (such as blindness, end-stage renal failure, liver cirrhosis, malignancy, chronic congestive heart failure)
* recent (within preceding 12 months) myocardial infarction, stroke or TIA
* unstable angina pectoris
* psychological conditions which may hamper patient's cooperation
* geographic inaccessibility
* any condition which, in the judgement of the Investigator, may make risky the participation in the study or bias the results

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of bariatric surgery in inducing partial or total remission of type 2 diabetes mellitus, as compared to standard medical anti-diabetic care (STC). | 10 years

SECONDARY OUTCOMES:
Secondary endpoints include percentage change of fasting plasma glucose levels, glycated hemoglobin, weight, waist circumference, blood pressure, cholesterol, HDL-cholesterol and triglycerides, hard cardiovascular risk and quality of life. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD, PhD, Principal Investigator — Catholic University Hospital; Giuseppe Nanni, MD, Study Chair — Catholic University Hospital
Locations (1):
- Catholic University, Faculty of Medicine, Rome, Italy

REFERENCES:
- [Background] Ferrannini E. Insulin resistance versus insulin deficiency in non-insulin-dependent diabetes mellitus: problems and prospects. Endocr Rev. 1998 Aug;19(4):477-90. doi: 10.1210/edrv.19.4.0336. PMID 9715376
- [Background] Weyer C, Tataranni PA, Bogardus C, Pratley RE. Insulin resistance and insulin secretory dysfunction are independent predictors of worsening of glucose tolerance during each stage of type 2 diabetes development. Diabetes Care. 2001 Jan;24(1):89-94. doi: 10.2337/diacare.24.1.89. PMID 11194248
- [Background] Ferrannini E, Gastaldelli A, Miyazaki Y, Matsuda M, Pettiti M, Natali A, Mari A, DeFronzo RA. Predominant role of reduced beta-cell sensitivity to glucose over insulin resistance in impaired glucose tolerance. Diabetologia. 2003 Sep;46(9):1211-9. doi: 10.1007/s00125-003-1169-6. Epub 2003 Jul 23. PMID 12879253
- [Background] Rossetti L, Giaccari A, DeFronzo RA. Glucose toxicity. Diabetes Care. 1990 Jun;13(6):610-30. doi: 10.2337/diacare.13.6.610. PMID 2192847
- [Background] Grill V, Bjorklund A. Dysfunctional insulin secretion in type 2 diabetes: role of metabolic abnormalities. Cell Mol Life Sci. 2000 Mar;57(3):429-40. doi: 10.1007/PL00000705. PMID 10823244
- [Background] Ferrannini E, Gastaldelli A, Miyazaki Y, Matsuda M, Mari A, DeFronzo RA. beta-Cell function in subjects spanning the range from normal glucose tolerance to overt diabetes: a new analysis. J Clin Endocrinol Metab. 2005 Jan;90(1):493-500. doi: 10.1210/jc.2004-1133. Epub 2004 Oct 13. PMID 15483086
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Ilkova H, Glaser B, Tunckale A, Bagriacik N, Cerasi E. Induction of long-term glycemic control in newly diagnosed type 2 diabetic patients by transient intensive insulin treatment. Diabetes Care. 1997 Sep;20(9):1353-6. doi: 10.2337/diacare.20.9.1353. PMID 9283777
- [Background] Karvestedt L, Andersson G, Efendic S, Grill V. A rapid increase in beta-cell function by multiple insulin injections in type 2 diabetic patients is not further enhanced by prolonging treatment. J Intern Med. 2002 Apr;251(4):307-16. doi: 10.1046/j.1365-2796.2002.00956.x. PMID 11952881
- [Background] Alvarsson M, Sundkvist G, Lager I, Henricsson M, Berntorp K, Fernqvist-Forbes E, Steen L, Westermark G, Westermark P, Orn T, Grill V. Beneficial effects of insulin versus sulphonylurea on insulin secretion and metabolic control in recently diagnosed type 2 diabetic patients. Diabetes Care. 2003 Aug;26(8):2231-7. doi: 10.2337/diacare.26.8.2231. PMID 12882841
- [Background] Ryan EA, Imes S, Wallace C. Short-term intensive insulin therapy in newly diagnosed type 2 diabetes. Diabetes Care. 2004 May;27(5):1028-32. doi: 10.2337/diacare.27.5.1028. PMID 15111515
- [Background] Salinari S, Bertuzzi A, Asnaghi S, Guidone C, Manco M, Mingrone G. First-phase insulin secretion restoration and differential response to glucose load depending on the route of administration in type 2 diabetic subjects after bariatric surgery. Diabetes Care. 2009 Mar;32(3):375-80. doi: 10.2337/dc08-1314. Epub 2008 Nov 25. PMID 19033407
- [Background] Cowan GS Jr, Buffington CK. Significant changes in blood pressure, glucose, and lipids with gastric bypass surgery. World J Surg. 1998 Sep;22(9):987-92. doi: 10.1007/s002689900504. PMID 9717426
- [Background] Marceau P, Hould FS, Simard S, Lebel S, Bourque RA, Potvin M, Biron S. Biliopancreatic diversion with duodenal switch. World J Surg. 1998 Sep;22(9):947-54. doi: 10.1007/s002689900498. PMID 9717420
- [Background] Scopinaro N, Adami GF, Marinari GM, Gianetta E, Traverso E, Friedman D, Camerini G, Baschieri G, Simonelli A. Biliopancreatic diversion. World J Surg. 1998 Sep;22(9):936-46. doi: 10.1007/s002689900497. PMID 9717419
- [Background] Greco AV, Mingrone G, Giancaterini A, Manco M, Morroni M, Cinti S, Granzotto M, Vettor R, Camastra S, Ferrannini E. Insulin resistance in morbid obesity: reversal with intramyocellular fat depletion. Diabetes. 2002 Jan;51(1):144-51. doi: 10.2337/diabetes.51.1.144. PMID 11756334
- [Background] Hickey MS, Pories WJ, MacDonald KG Jr, Cory KA, Dohm GL, Swanson MS, Israel RG, Barakat HA, Considine RV, Caro JF, Houmard JA. A new paradigm for type 2 diabetes mellitus: could it be a disease of the foregut? Ann Surg. 1998 May;227(5):637-43; discussion 643-4. doi: 10.1097/00000658-199805000-00004. PMID 9605655
- [Background] Mari A, Manco M, Guidone C, Nanni G, Castagneto M, Mingrone G, Ferrannini E. Restoration of normal glucose tolerance in severely obese patients after bilio-pancreatic diversion: role of insulin sensitivity and beta cell function. Diabetologia. 2006 Sep;49(9):2136-43. doi: 10.1007/s00125-006-0337-x. Epub 2006 Jul 4. PMID 16819611
- [Background] Muscelli E, Mingrone G, Camastra S, Manco M, Pereira JA, Pareja JC, Ferrannini E. Differential effect of weight loss on insulin resistance in surgically treated obese patients. Am J Med. 2005 Jan;118(1):51-7. doi: 10.1016/j.amjmed.2004.08.017. PMID 15639210
- [Background] Rubino F, Gagner M, Gentileschi P, Kini S, Fukuyama S, Feng J, Diamond E. The early effect of the Roux-en-Y gastric bypass on hormones involved in body weight regulation and glucose metabolism. Ann Surg. 2004 Aug;240(2):236-42. doi: 10.1097/01.sla.0000133117.12646.48. PMID 15273546
- [Background] Naslund E, Backman L, Holst JJ, Theodorsson E, Hellstrom PM. Importance of small bowel peptides for the improved glucose metabolism 20 years after jejunoileal bypass for obesity. Obes Surg. 1998 Jun;8(3):253-60. doi: 10.1381/096089298765554449. PMID 9678192
- [Background] le Roux CW, Aylwin SJ, Batterham RL, Borg CM, Coyle F, Prasad V, Shurey S, Ghatei MA, Patel AG, Bloom SR. Gut hormone profiles following bariatric surgery favor an anorectic state, facilitate weight loss, and improve metabolic parameters. Ann Surg. 2006 Jan;243(1):108-14. doi: 10.1097/01.sla.0000183349.16877.84. PMID 16371744
- [Background] Clements RH, Gonzalez QH, Long CI, Wittert G, Laws HL. Hormonal changes after Roux-en Y gastric bypass for morbid obesity and the control of type-II diabetes mellitus. Am Surg. 2004 Jan;70(1):1-4; discussion 4-5. PMID 14964537
- [Background] Lauritsen KB, Christensen KC, Stokholm KH. Gastric inhibitory polypeptide (GIP) release and incretin effect after oral glucose in obesity and after jejunoileal bypass. Scand J Gastroenterol. 1980;15(4):489-95. doi: 10.3109/00365528009181506. PMID 7001614
- [Background] Rubino F, Marescaux J. Effect of duodenal-jejunal exclusion in a non-obese animal model of type 2 diabetes: a new perspective for an old disease. Ann Surg. 2004 Jan;239(1):1-11. doi: 10.1097/01.sla.0000102989.54824.fc. PMID 14685093
- [Background] Sirinek KR, O'Dorisio TM, Hill D, McFee AS. Hyperinsulinism, glucose-dependent insulinotropic polypeptide, and the enteroinsular axis in morbidly obese patients before and after gastric bypass. Surgery. 1986 Oct;100(4):781-7. PMID 3532392
- [Background] Morinigo R, Moize V, Musri M, Lacy AM, Navarro S, Marin JL, Delgado S, Casamitjana R, Vidal J. Glucagon-like peptide-1, peptide YY, hunger, and satiety after gastric bypass surgery in morbidly obese subjects. J Clin Endocrinol Metab. 2006 May;91(5):1735-40. doi: 10.1210/jc.2005-0904. Epub 2006 Feb 14. PMID 16478824
- [Background] Valverde I, Puente J, Martin-Duce A, Molina L, Lozano O, Sancho V, Malaisse WJ, Villanueva-Penacarrillo ML. Changes in glucagon-like peptide-1 (GLP-1) secretion after biliopancreatic diversion or vertical banded gastroplasty in obese subjects. Obes Surg. 2005 Mar;15(3):387-97. doi: 10.1381/0960892053576613. PMID 15826475
- [Background] Jorde R, Burhol PG, Johnson JA. The effect of jejunoileal bypass on postprandial release of plasma gastric inhibitory polypeptide (GIP). Scand J Gastroenterol. 1981;16(2):313-9. doi: 10.3109/00365528109181974. PMID 7031848
- [Background] Sarson DL, Scopinaro N, Bloom SR. Gut hormone changes after jejunoileal (JIB) or biliopancreatic (BPB) bypass surgery for morbid obesity. Int J Obes. 1981;5(5):471-80. PMID 6796532
- [Derived] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Capristo E, Chamseddine G, Bornstein SR, Rubino F. Metabolic surgery versus conventional medical therapy in patients with type 2 diabetes: 10-year follow-up of an open-label, single-centre, randomised controlled trial. Lancet. 2021 Jan 23;397(10271):293-304. doi: 10.1016/S0140-6736(20)32649-0. PMID 33485454
- [Derived] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Nanni G, Castagneto M, Bornstein S, Rubino F. Bariatric-metabolic surgery versus conventional medical treatment in obese patients with type 2 diabetes: 5 year follow-up of an open-label, single-centre, randomised controlled trial. Lancet. 2015 Sep 5;386(9997):964-73. doi: 10.1016/S0140-6736(15)00075-6. PMID 26369473
- [Derived] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317